CLINICAL TRIAL: NCT00087880
Title: Maintaining Abstinence in Chronic Cigarette Smokers
Brief Title: Maintaining Abstinence in Chronic Cigarette Smokers - 1
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: National Institute on Drug Abuse (NIDA) (NIH)
Responsible Party: Sharon M. Hall, Ph.D, University California, San Francisco
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: NIDA-15732-1; R01-15732-1
Record Dates: First submitted 2004-07-15; First posted 2004-07-19 (Estimated); Last update posted 2017-01-12 (Estimated); Status verified 2016-03

CONDITIONS: Tobacco Use Disorder
Keywords: smoking cessation
MeSH Terms: conditions — Tobacco Use Disorder; Smoking Cessation | interventions — Bupropion; Nicotine Replacement Therapy

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (5):
- Brief Treatment (Active Comparator): Participants will start with a 21 mg nicotine patch, tapering to 14 mg patch and finally tapering to 7 mg patch. The nicotine patch will be administered on Week 3 of the program. Participants will meet with medical staff during Weeks 1, 2, 5, and 11. Five group counseling sessions must be attended by the participants. Assessments will be conducted on Weeks 12, 24, 36, 52, 64, and 104.
  Interventions: Drug: Bupropion and NRT
- Extended Bupropion/Low Contact (Active Comparator): Participants will receive the Brief Treatment followed by ongoing Bupropion treatment through Week 52. Participants will meet with medical staff once a month.
  Interventions: Drug: Bupropion and NRT
- Extended Placebo/Low Contact (Placebo Comparator): Participants will receive the Brief Treatment followed by placebo medication (sugar-pill) through Week 52 and meet with medical staff once a month.
  Interventions: Drug: Bupropion and NRT
- Extended Bupropion/High Contact (Active Comparator): Participants will receive Brief Treatment followed by ongoing bupropion treatment through Week 52. Participants will attending counseling session 20-40 minutes in duration and will be scheduled at weeks 12, 14, 16, 18, 20, 24, 28, 32, 36, 44, and 52. The contents of these sessions will introduce additional information focusing on motivation, social support, mood management, weight gain, and dependence/withdrawal. Subjects will be contact by phone between counseling sessions (at Weeks 13, 15, 18, 22, 26, 30, 34, 36, 40, 48) for a brief check-in.
  Interventions: Drug: Bupropion and NRT
- Extended Placebo/High Contact (Placebo Comparator): Participants receive the Brief Treatment followed by a placebo medication through Week 52 and meet with medical staff once per month. Participants will attending counseling session 20-40 minutes in duration and will be scheduled at weeks 12, 14, 16, 18, 20, 24, 28, 32, 36, 44, and 52. The contents of these sessions will introduce additional information focusing on motivation, social support, mood management, weight gain, and dependence/withdrawal. Subjects will be contact by phone between counseling sessions (at Weeks 13, 15, 18, 22, 26, 30, 34, 36, 40, 48) for a brief check-in.
  Interventions: Drug: Bupropion and NRT

INTERVENTIONS:
Drug: Bupropion and NRT — All participants receive standard 12 week treatment of NRT, bupropion and five group counseling sessions. At week 11, subjects are randomly assigned to one of five treatment groups (1) Bupropion/Low Contact; (2) Placebo/Low Contact; (3) Bupropion/Relapse Prevention; (4) Placebo/Relapse Prevention; (5) No Further Treatment. Data is collected at Week 0, and at weeks 12, 24, 52, 64, and 104.
  Other Names: Zyban

SUMMARY:
The purpose of this study is to evaluate the extended pharmacological and psychological treatment for chronic cigarette smokers.

DETAILED DESCRIPTION:
The work adapts interventions that have been successful in the general populations, and tailors them to chronic smokers, who may have numerous previous smoking treatment failures. If successful it will: (1) make available a treatment intervention that produces hight long term abstinence rates; (2) provide information on variables that predicts success and failure in this population of smokers; (3) examine the cost-effectiveness of more intensive, longer term treatments.

ELIGIBILITY:
Subjects (N=400) will be men and women (50%) over the age of 18 who smoke at least 10 cigarettes per day and answers yes to the question "Do you smoke within 30 minutes of arising?"

Inclusion Criteria:

-Subjects are age 18 and over, currently smoking 10 or more cigarettes per day, and report a smoking history of at least 5 years in response to the question "How long have you been a regular smoker?"

Exclusion Criteria:

* History of seizure or head injury resulting in unconsciousness
* Any condition that might predispose to seizures (brain tumor or stroke)
* A current or history of anorexia nervosa or bulimia
* Any disease acutely life-threatening or so severe that the patient is judged unable to comply with the protocol
* Use of a protease inhibitor of MAO inhibitor within the last two week
* Current use of psychiatric drugs that would interfere with interpretation of study results, including antidepressants
* Treatment for alcohol dependence during the last year, or evidence of alcohol abuse so severe that the patient is judged potentially unable to comply with the protocol
* Patients who know they are leaving the Bay Area within the study period and non-English speakers will be excluded
* Suicidal or homicidal ideation
* Current major depression
* History of bipolar disorder
* Recent (within twelve months) myocardial infarction
* Any other medical condition that would contraindicate use of NRT or bupropion
* Physical limitation so severe that participation in a program of moderate exercise is not possible
* Pregnancy or lactation

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 407 (Actual)
Dates: Start 2002-12; Primary Completion 2005-01 (Actual); Study Completion 2009-09 (Actual)

PRIMARY OUTCOMES:
Smoking Behavior | 2

CONTACTS AND LOCATIONS:
Overall Officials: Sharon M Hall, Ph.D., Principal Investigator — University of California, San Francisco
Locations (1):
- University California, San Francisco, San Francisco, California, United States

REFERENCES:
- [Derived] Hajizadeh A, Howes S, Theodoulou A, Klemperer E, Hartmann-Boyce J, Livingstone-Banks J, Lindson N. Antidepressants for smoking cessation. Cochrane Database Syst Rev. 2023 May 24;5(5):CD000031. doi: 10.1002/14651858.CD000031.pub6. PMID 37230961